CLINICAL TRIAL: NCT02445079
Title: Epidemiology of Atherosclerosis Among Older-Age People in Southwestern Uganda
Brief Title: Ugandan Non-Communicable Diseases and Aging Cohort
Acronym: UGANDAC
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Mbarara University of Science and Technology (Other); University of California, San Francisco (Other); Ragon Institute of MGH, MIT and Harvard (Other); National Institutes of Health (NIH) (NIH); Harvard University (Other)
Responsible Party: Principal Investigator, Mark Siedner, Assistant in Medicine, Massachusetts General Hospital
Other Study IDs: 2014P001928
Record Dates: First submitted 2015-05-06; First posted 2015-05-15 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: HIV; Cardiovascular Disease; Chronic Obstructive Pulmonary Disease; Atherosclerosis; Hypertension; Diabetes Mellitus
MeSH Terms: conditions — Cardiovascular Diseases; Pulmonary Disease, Chronic Obstructive; Atherosclerosis; Hypertension; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Annual collection of serum, plasma, and stool.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HIV infected: HIV infected sub-group
  Interventions: Other: This is an observational study only
- HIV uninfected: HIV uninfected sub-group, age and gender matched to the HIV-infected group
  Interventions: Other: This is an observational study only

INTERVENTIONS:
Other: This is an observational study only — Observational study only

SUMMARY:
Longitudinal cohort study of older-aged people living with HIV infection in southwestern Uganda and age and gender-matched HIV uninfected controls with the primary aim of measuring the epidemiology of cardiovascular and pulmonary disease in this study setting, and particularly the contribution of HIV infection to it.

DETAILED DESCRIPTION:
This study recruits people living with HIV/AIDS (PLWH) aged 40 and older; and an HIV-uninfected age and gender-matched, community-based comparison group in the HIV clinic catchment area.

Study investigators will collect sociodemographic, clinical, immune activation, systemic inflammation, plasma and stool microbiome, and clinical pulmonary and cardiovascular disease measures. Our outcomes of interest are measures of carotid atherosclerosis, including carotid intima media thickness and presence of plaque, prior ischemic heart disease (as measured by electrocardiograms), peripheral arterial disease (as measured by ankle-branchial index), and lung function as measured by pulmonary function testing. Our exposures of interest are traditional cardiovascular disease risk factors (e.g. age, gender, family history of cardiovascular disease, smoking history, diet, activity, body mass index, prevalence of diabetes, and prevalence of hypertension) and HIV-related cardiovascular risk factors (e.g. nadir CD4 count, ART duration and regimen, gut and plasma microbiome composition, and markers of both immune activation and systemic inflammation).

Investigators will collect this data to accomplish the following aims:

Aim 1: Compare the prevalence of atherosclerosis, measured by cIMT, ankle-brachial index, and presence of q-waves on electrocardiogram, in PLWH taking ART aged 40 and older and age and gender-matched, population-based HIV-uninfected controls. This study aims to be among the first to capture high-quality measures of atherosclerotic disease among a population of PLWH in sub-Saharan Africa. The study aims to test the hypothesis that older-age Ugandans on ART will have thicker carotid intima media, higher prevalence of peripheral arterial disease, and higher prevalence of pathologic q-waves on electrocardiogram than age and gender-matched, HIV-uninfected controls.

Aim 2: Evaluate correlates of atherosclerosis in older-age PLWH on ART, including both traditional (age, gender, smoking, diabetes and hypertension prevalence) and HIV-related risk factors (immune activation, systemic inflammation, and stool and plasma microbiome composition). The study will leverage a collaboration with the Ragon Institute to perform immunologic and molecular testing for microbial translocation and markers of immune activation and systemic inflammation (e.g. soluble CD163, C-reactive protein, IL-6, CD8+ T-lymphocyte activation).

Aim 3: Compare the progression of atherosclerosis in PLWH versus HIV-uninfected individuals over five years of observation time. The study aims to test the hypothesis that the rate of change in carotid intima media thickness will be faster in among PLWH over 45 on ART than age and gender-matched HIV-uninfected controls, and that rates of change in carotid intima media thickness among the HIV-infected cohort will be associated with markers of microbial translocation, immune activation, and systemic inflammation.

Aim 4: Compare the prevalence and incidence of abnormal pulmonary function (FEV1, FVC, FEV1/FVC) in PLWH on ART and age- and gender-matched, population-based HIV-uninfected controls, utilizing handheld spirometry with bronchodilator challenge. The study aims to test the hypothesis that pulmonary function is worse and COPD is more common among people living with HIV/AIDS than age- and gender-match HIV-uninfected controls.

ELIGIBILITY:
Group 1 Inclusion Criteria:

* HIV infected
* Age > 40 years old at enrollment
* Minimum 2 years of antiretroviral therapy

Group 1 Exclusion Criteria:

* Decline informed consent

Group 2 Inclusion Criteria:

* Living in catchment area of Mbarara Regional Referral Hospital (greater Mbarara)
* Age > 40 years old
* Age and gender matched to a participant in group 1

Group 2 Exclusion Criteria:

* HIV infection (tested annually as part of study procedures)
* Decline informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study recruits two sub-groups of participants:
  Study Group 1:
  -HIV infected persons aged 40 and older, in care at the Immune Suppression Syndrome HIV Clinic at Mbarara Regional Referral Hospital
  Study Group 2:
  -Community-based, HIV uninfected persons recruited from the catchment area of the Mbarara Regional Referral Hospital (greater Mbarara), and age and gender-matched to Group 1 participants
Sampling Method: Non-Probability Sample
Enrollment: 309 (Actual)
Dates: Start 2013-12; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Baseline prevalence and incident change in carotid intima media thickness | Outcomes will be collected at baseline and every 12 months (i.e. months 12, 24, 36, 48, and 60) for study duration (planned 60 months)
  Measured by carotid ultrasonography

SECONDARY OUTCOMES:
Baseline prevalence and incident change in carotid plaque | Outcomes will be collected at baseline and every 12 months (i.e. months 12, 24, 36, 48, and 60) for study duration (planned 60 months)
  Measured by carotid ultrasonography
Baseline prevalence and incident change in ischemic heart disease | Outcomes will be collected at baseline and every 12 months (i.e. months 12, 24, 36, 48, and 60) for study duration (planned 60 months)
  Measured by electrocardiography
Baseline prevalence and incident change in peripheral arterial disease | Outcomes will be collected at baseline and every 12 months (i.e. months 12, 24, 36, 48, and 60) for study duration (planned 60 months)
  Measured by ankle branchial index
Baseline prevalence and incident change in chronic obstructive pulmonary disease | Outcomes will be collected at baseline and every 12 months (i.e. months 12, 24, 36, 48, and 60) for study duration (planned 60 months)
  Measured by pulmonary function testing

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Siedner, MD MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Mbarara University of Science and Technology, Mbarara, Uganda

REFERENCES:
- [Derived] Siedner MJ, Bibangambah P, Kim JH, Lankowski A, Chang JL, Yang IT, Kwon DS, North CM, Triant VA, Longenecker C, Ghoshhajra B, Peck RN, Sentongo RN, Gilbert R, Kakuhikire B, Boum Y 2nd, Haberer JE, Martin JN, Tracy R, Hunt PW, Bangsberg DR, Tsai AC, Hemphill LC, Okello S. Treated HIV Infection and Progression of Carotid Atherosclerosis in Rural Uganda: A Prospective Observational Cohort Study. J Am Heart Assoc. 2021 Jun 15;10(12):e019994. doi: 10.1161/JAHA.120.019994. Epub 2021 Jun 5. PMID 34096320